CLINICAL TRIAL: NCT02165384
Title: Continued Evaluation of the Preceptis Medical, Inc. Tympanostomy Ear Tube Introducer
Brief Title: Hummingbird TTS Ear Tube Delivery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Preceptis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Preceptis Alpha
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Otitis Media
Keywords: tympanostomy; myringotomy; otitis media; ear tubes; ear infection
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hummingbird TTS (Experimental): Ear tube placement with the Hummingbird TTS
  Interventions: Device: Ear tube placement with the Hummingbird TTS

INTERVENTIONS:
Device: Ear tube placement with the Hummingbird TTS — Using the Hummingbird TTS to make a myringotomy and deliver a tympanostomy tube across the tympanic membrane with one pass.
  Other Names: Preceptis Medical, Inc. Tympanostomy Tube Introducer System; Hummingbird Tympanostomy Tube Delivery System; Hummingbird TTS

SUMMARY:
The purpose of this study is to determine if the Hummingbird ear tube delivery system is a safe and effective way to put ear tubes in place.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and performance of the TTI device for the placement of ear tubes in patients undergoing a tympanostomy tube placement procedure.The trial will be a multi-site, prospective, treatment only study of the Preceptis ear tube introducer . Patients will already have a scheduled tympanostomy procedure. Enrollment in the study at each site will begin after receipt of Institutional Review Board (IRB) approval. Patients will be considered enrolled at the time the informed consent document is signed. A maximum of two hundred fifty (250) subjects will be included in the study at up to 5 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo tympanostomy tube insertion.
2. At least 6 months old.
3. Subject is able and willing to comply with follow-up requirements.
4. Signed Informed Consent, Parental Consent Form, or Child Assent Form as applicable.

Exclusion Criteria:

1. Any condition that in the opinion of the investigator may place the subject at greater risk (e.g., pregnancy)
2. Significantly atrophic tympanic membrane.
3. Significantly atelectatic tympanic membrane. For example, the tympanic membrane is in contact with the promontory of the cochlea.
4. Anatomy precludes sufficient visualization and access to the tympanic membrane.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Rimell, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (4):
- United States (4):
  - Fairview Maple Grove Surgery Center, Maple Grove, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Hummingbird TTS: Treatment only surgical instrument study
Period: Overall Study
Arm/Group | Hummingbird TTS
Started | 199
Completed | 199
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients scheduled for tympanostomy tube insertion that are at least 6 months old
Arm/Group | Hummingbird TTS
Number analyzed (Participants) | 199
Age, Customized [Median (Full Range); unit: months] | 20 [6 to 182]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender not important or captured for this study
  Male | NA — Gender not important or captured for this study
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race not captured
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 199
Region of Enrollment [Number; unit: participants]
  United States | 199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ears in Which an Ear Tube Was Successfully Delivered Across the Tympanic Membrane
Description: Success will be determined at the end of each ear tube procedure, by whether or not the TTS was used during the tympanostomy procedure to make an incision in the tympanic membrane and deploy an ear tube. Data may be presented when enrollment has been completed and all pre-operative and procedure data are analyzed.
Time Frame: intra operative
Population: 393 ears in 199 patients received ear tube placement from the Hummingbird device.
Measure: Count of Units; unit: Ears
Units Other Than Participants: Ears
Groups:
- Hummingbird TTS: Treatment only HTTS was used to make incision and deliver ear tube
Arm/Group | Hummingbird TTS
Number analyzed (Participants) | 199
Number analyzed (Ears) | 393
Ears | 393

2. Primary Outcome: Number of Participants With Intra-operative Adverse Events
Description: Any intra-operative adverse events, anticipated or unanticipated
Time Frame: Intra-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Hummingbird TTS
Number analyzed (Participants) | 199
Participants | 0

ADVERSE EVENTS:
Time Frame: Intra-operative
Arm/Group | Hummingbird TTS
All-Cause Mortality (participants affected / at risk) | 0/199
Serious Adverse Events (participants affected / at risk) | 0/199
Other Adverse Events (participants affected / at risk) | 0/199

LIMITATIONS AND CAVEATS:
Non-significant risk study. Treatment only evaluation of a surgical instrument used for tympanostomy procedures.

Other instruments could be used during the tympanostomy procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT02165384/Prot_SAP_000.pdf